CLINICAL TRIAL: NCT06966596
Title: Effect of Low-Dose Ketamine Infusion on Quality and Duration of Post-Operative Pain in Patients Undergoing Laparoscopic Cholecyctectomy Under General Anesthesia
Brief Title: Low-Dose Ketamine Infusion for Post-Operative Pain in Patients Undergoing Laparoscopic Cholecyctectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fazaia Ruth Pfau Medical College (Other)
Responsible Party: Principal Investigator, Syeda Hajrah Rehman, Principal Investigator, Fazaia Ruth Pfau Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FPRMC-IRB-2024-38
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Cholelithiasis; Cholecystectomy; Laparoscopic surgery; Ketamine; Analgesia
MeSH Terms: conditions — Cholelithiasis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A received ketamineat 0.2mg/kg bolus intravenously followed by ketamine infusion at rate of 0. (Experimental): Group A received ketamineat 0.2mg/kg bolus intravenously followed by ketamine infusion at rate of 0.2mg/kg/hr throughout the surgery.
  Interventions: Drug: Ketamine only
- Control Group B (Placebo Comparator): Control group received normal saline intravenously at an equivalent infusion rate
  Interventions: Other: Placebo Normal Saline (NS)

INTERVENTIONS:
Drug: Ketamine only — Group A received ketamineat 0.2mg/kg bolus intravenously followed by ketamine infusion at rate of 0.2mg/kg/hr throughout the surgery. W
  Arms: Group A received ketamineat 0.2mg/kg bolus intravenously followed by ketamine infusion at rate of 0.
Other: Placebo Normal Saline (NS) — Control group received normal saline to maintain double blinding
  Arms: Control Group B

SUMMARY:
Following surgery, acute pain is a typical issue with a variety of implications. Surgeons, anesthesia specialists, and patients all desire effective pain management with the fewest possible adverse effects. At low dosages (<0.3 mg/kg/hr) and large doses (>1 mg/kg), ketamine is utilized as an analgesic and an anaesthetic. Ketamine at high dosages causes dissociative anaesthesia with little impact on breathing or airway reflexes. Although this medication is a powerful analgesic, its usage is restricted due to it leads to agitation and hallucinations during awakening. Nevertheless, it has a potent analgesic effect when administered at a subanesthetic dose, and ketamine's psychomimetic side effects are rare at these dosages. This study intended to examine the role of low-dose for post-operative pain control in patients undergoing LC, despite the fact that numerous studies have been conducted on the subject and that the results have been inconsistent.

DETAILED DESCRIPTION:
Most patients still stay overnight after a laparoscopic cholecystectomy (LC) due to post-operative pain, which continues to be the principal obstacle to early patient discharge. On the first postoperative day following laparoscopic procedures, patients may have mild to moderate postoperative pain, with decreased pain intensity in the shoulder area (from the subdiaphragmatic region), particularly intra-abdominal and local discomfort at the incision site. Because of its analgesic properties and cardiovascular stability, ketamine has been used extensively in anesthesia practice. It non-competitively blocks N-methyl-D-aspartate (NMDA) receptors. As an addition to multimodal perioperative pain management, ketamine has grown in favor in recent years. Ketamine at high dosages causes dissociative anaesthesia with little impact on breathing or airway reflexes. In a range of surgical procedures, low-dose ketamine infusions (<0.3 mg/kg/hr) have demonstrated effectiveness in lowering pain scores and minimising the need for postoperative opioids. Regarding the reduction of pain and analgesic demand, ketamine has demonstrated conflicting effects. The study objective was to determine the effect of low-dose ketamine infusion on quality and duration of post-operative pain in patients undergoing laparoscopic in a tertiary care hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 18 years or above of either gender
* Patients planned of elective laparoscopic choleycyctectomy

Exclusion Criteria:

* Obese patients
* History of alcohol consumption and drug abusers
* Uncontrolled hypertension
* Uncontrolled diabetes
* Patients with chronic pain
* Patients allergic to study drugs
* Patients with neurological disorders
* Patients unable to understand scoring system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Post-pain assessment | pain status was monitored post-operatively at 0 hour, 2 hour, 4 hours, 6 hours, 12 hours and at 24 hours
  pain was assessed using numeric rating scale which is a ten point scoring scale ranging from 0-10 for ranking pain where 0 means no pain and 10 means worst pain.

SECONDARY OUTCOMES:
time to rescue analgesia | till 24 hours post-operatively
  time to rescue analgesia was defined as time point at which patient was given rescue analgesia for pain score of 5 or above

CONTACTS AND LOCATIONS:
Locations (1):
- Fazaia Ruth Pfau Medical College, PAF Hospital Base Faisal, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
This is institutional data which has to be concealed for patient's privacy

REFERENCES:
- [Background] Jain S, Nazir N, Mustafi SM. Preemptive low-dose intravenous ketamine in the management of acute and chronic postoperative pain following laparoscopic cholecystectomy: a prospective randomized control study. Med Gas Res. 2022 Oct-Dec;12(4):141-145. doi: 10.4103/2045-9912.337995. PMID 35435425
- [Background] Akturk R, Serinsoz S. Determining a Method to Minimize Pain After Laparoscopic Cholecystectomy Surgery. Surg Laparosc Endosc Percutan Tech. 2022 Aug 1;32(4):441-448. doi: 10.1097/SLE.0000000000001071. PMID 35797664
- [Background] Gin E, Lowen D, Tacey M, Hodgson R. Reduced Laparoscopic Intra-abdominal Pressure During Laparoscopic Cholecystectomy and Its Effect on Post-operative Pain: a Double-Blinded Randomised Control Trial. J Gastrointest Surg. 2021 Nov;25(11):2806-2813. doi: 10.1007/s11605-021-04919-0. Epub 2021 Feb 9. PMID 33565010